CLINICAL TRIAL: NCT00681031
Title: An Open-label, Single-arm, Phase IV Study Assessing the Immunogenicity and Safety of ZOSTAVAX® at Minimum Release Specification Approaching Expiry Potency in Subjects ≥50 Years Old.
Brief Title: Zostavax® at Minimum Release Specification Approaching Expiry (V211-044)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V211-044; ZTV02C (Other: MCMVaccBV (SPMSD) Protocol Number); 2007-006532-66 (EudraCT Number)
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Enrolled (Experimental): Participants received a single dose (0.65 mL) of shingles (herpes zoster) vaccine (live) ZOSTAVAX® by subcutaneous injection at Visit 1 (Day 0)
  Interventions: Biological: ZOSTAVAX®

INTERVENTIONS:
Biological: ZOSTAVAX® — One dose (0.65 mL) contains: Varicella-zoster virus, Oka/Merck strain, (live attenuated) not less than 19400 PFU

SUMMARY:
Primary objective:

To demonstrate whether or not ZOSTAVAX® at minimum release specification approaching expiry potency elicits an acceptable Varicella-Zoster Virus (VZV) antibody fold rise (measured by glycoprotein Enzyme Linked ImmunoSorbent Assay [gpELISA]) from pre-vaccination to 4 weeks post-vaccination.

Secondary objectives:

To describe the safety profile of ZOSTAVAX® at minimum release specification approaching expiry potency.

ELIGIBILITY:
Inclusion Criteria:

* Participant of either gender aged ≥50 years
* Positive history of varicella or residence for >30 years in a country with endemic VZV infection
* All females must be postmenopausal or have a negative serum or urine pregnancy test or acceptable method of birth control for three months after vaccination
* Participant having signed the informed consent form prior to any study procedure

Exclusion Criteria:

* Febrile within 72 hours prior to vaccination
* Prior history of Herpes Zoster clinically diagnosed by a physician
* Previously received a varicella or zoster vaccine
* Exposure to varicella or herpes-zoster within 4 weeks prior to vaccination
* Received any other live virus vaccine within 4 weeks prior to vaccination, or is expected to receive any other live virus vaccine during the study
* Received any inactivated vaccine within 2 weeks prior to vaccination, or is expected to receive any inactivated vaccine during the study
* Was treated with immunoglobulins or any blood products, other than autologous blood transfusion, given during the 5 months prior to vaccination or is expected to be treated during the study
* Taking any non topical antiviral therapy with activity against herpesviruses.
* On immunosuppressive therapy
* Known or suspected immune dysfunction caused by a medical condition, or any other cause
* History of hypersensitivity reaction or anaphylactoid reaction to any vaccine component, including gelatin or neomycin
* Known active tuberculosis
* Significant underlying illness preventing completion of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-05-14 (Actual); Primary Completion 2008-06-25 (Actual); Study Completion 2008-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Arnou R, Fiquet A, Thomas S, Sadorge C. Immunogenicity and safety of ZOSTAVAX((R)) approaching expiry potency in individuals aged >/=50 years. Hum Vaccin. 2011 Oct;7(10):1060-5. doi: 10.4161/hv.7.10.16480. Epub 2011 Oct 1. PMID 21941091

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Enrolled
Started | 96
Completed | 96
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 46

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titre (GMT) of Varicella Antibodies
Description: Blood samples to determine the GMT of varicella antibodies taken pre-vaccination and again 28 to 35 days post vaccination. Titres determined by glycoprotein enzyme-linked immunosorbent assay (gpELISA).
Time Frame: Predose (Day 0) and Day 28-35 Post Dose
Population: All vaccinated participants excluding those with any protocol deviation which may have interfered with the immunogenicity evaluation and excluding participants with herpes zoster onset before the post-vaccination blood sample
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | All Enrolled
Number analyzed (Participants) | 92
gpELISA units/mL
  Predose | 215.8 [178.1 to 261.4]
  Postdose | 674.0 [565.4 to 803.5]
Statistical Analysis 1: Comparison: All Enrolled; Test type: Non-Inferiority or Equivalence — Acceptability was demonstrated if the lower bound of the two-sided 95% confidence interval (CI) on the Geometric Mean Fold Rise (CMFR) from pre-vaccination to 4 weeks postvaccination is >1.4; GMFR = 3.1, 95% CI 2-sided [2.6 to 3.8] — GMFR = GMT postdose divided by GMT predose

ADVERSE EVENTS:
Time Frame: Up to 35 days post vaccination
Groups:
- V211: All enrolled participants who received vaccination
Arm/Group | V211
Serious Adverse Events (participants affected / at risk) | 0/96
Other Adverse Events (participants affected / at risk) | 50/96
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V211 (N=96)
Injection site erythema (General disorders) | 36 (36)
Injection site pain (General disorders) | 39 (39)
Injection site swelling (General disorders) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall send to Sanofi Pasteur MSD for approval any of the publication and/or communication draft, in whatever forms (abstracts, manuscripts, texts). Sanofi Pasteur MSD shall have 60 (sixty) days to review the draft, have reserves if any, and formulate its refusal to the draft in whole or in part if the draft contains confidential data, may prejudice to Sanofi Pasteur MSD patent/intellectual property rights and/or is not compliant with the study results.